CLINICAL TRIAL: NCT02467296
Title: Rationale and Design of the PRevent Adverse Outcomes in Heart faIlure By limITing Sodium Study
Brief Title: Dietary Sodium Intake and Outcomes in Heart Failure
Acronym: PROHIBITSodium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Javed Butler, MD, MPH, MBA, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1R34HL119773 (NIH); 639316 (Other: Stony Brook CORIHS A); R34HL119773 (NIH)
Record Dates: First submitted 2015-06-03; First posted 2015-06-10 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Heart Failure
Keywords: Sodium; outcomes
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: 1.5 gr of Sodium (Active Comparator): Meal Plans with 1.5 gr of Sodium
  Interventions: Other: Dietary plan with controlled amount of Sodium
- B: 3 gr of Sodium (Active Comparator): Meal Plans with 3 gr of Sodium
  Interventions: Other: Dietary plan with controlled amount of Sodium

INTERVENTIONS:
Other: Dietary plan with controlled amount of Sodium — Dietary plan with 1.5 gr vs 3 gr of Sodium

SUMMARY:
Currently, the recommendations for sodium intake restriction for patients with heart failure are mostly based on expert consensus and observational evidence, whereas smaller randomized studies have actually suggested that strict dietary sodium reduction may be harmful in heart failure. In the present clinical trial pilot study, the investigators plan to collect data on enrollment rates, compliance, outcomes, and safety of a 12-week dietary intervention in heart failure patients, with prepared food containing two different levels of sodium (1,500 mg and 3,000 mg) daily, followed by a 12-week surveillance for safety and effectiveness. The goal is to inform the design of a fullscale clinical trial that will provide more definitive evidence for dietary sodium recommendations in heart failure.

DETAILED DESCRIPTION:
Despite the intense research for improving outcomes in heart failure, evidence remains scarce (and mostly observational) for dietary sodium restriction, arguably the most widely recommended self-care measure for heart failure. In explicit acknowledgement of the evidence gaps and unclear benefits, the recent European Society of Cardiology guidelines have not assigned a level of evidence to sodium intake recommendations and the American College of Cardiology (ACC) and American Heart Association (AHA) guidelines do not provide a specific target level of sodium intake for patients with HF.

Although it seems reasonable to restrict sodium below <3000 mg/d in heart failure, it is currently unknown how "low" is appropriate for these patients.

This study will attempt to provide the basis to evaluate the above guidelines by determining, in consecutive HFrEF patients with EF ≤40% during an acute HF admission, the proportion of patients who: (1) are willing to participate in a 12-week feeding trial; (2) meet the trial eligibility criteria; and (C) subsequently continue to consume ≥3000 mg/d sodium 15-30 days post discharge despite discharge instructions. This will allow the investigators to estimate enrollment rates in a full-scale trial.

This study will randomize 50 eligible patients to prepared meal plans with either 1500 mg/d vs. 3000 mg/d sodium for 12 weeks .

The hypotheses of the present study are that (1) ≥ 90% of patients will be retained on the study by 12 weeks (or at first outcome or safety event) and (2) patients will be compliant with provided food ≥ 90% of the study days.

Study Primary Endpoints:

(i) Overall on-study retention and (ii) compliance with the prepared food, assessed via daily food diaries and 24-h urine collections at baseline, 4, 8, and 12 weeks.

Study Secondary Endpoints:

Estimate trends in (1) all-cause mortality, readmissions, and emergency room visits; (2) NT-pro-B-type natriuretic peptide levels; and (3) diet palatability and quality of life, between the two arms.

Safety endpoints:

Safety of the intervention assessed by vital sign and laboratory assessments. This pilot study is expected to yield critical information necessary and sufficient to design a full-scale clinical trial that will provide evidence for dietary sodium recommendations in heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥21 years at screening
2. Recent (≤1 year) EF ≤40%
3. Standard HF treatment, including ACEI/ARB & beta-blockers & aldosterone antagonists, unless contraindicated or intolerant

5. Able to consume research diet (e.g. no dysphagia etc.) 6. Systolic blood pressure ≥100 mmHg 7. >3000 mg/d sodium excretion (by 24-hr urinary sodium)

Exclusion Criteria:

1. Institutionalized patients
2. Siogns or symptoms of instability in HF status
3. Communication barriers, including cognitive impairment; inability to communicate and understand and cooperate with the protocol
4. Severe non-cardiac illness that compromises life expectancy within the next 12 months or the ability to participate in the study (e.g. severe hepatobiliary disease, cancer underground chemo- or radiotherapy)
5. Any medical or surgical procedure planned in the next 6 months
6. Participants planning to move to a different state within 6 months
7. Participation in any other experimental protocol
8. Renal replacement therapy or Stage 4 or 5 chronic kidney disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Patient On-Study Retention | 3 month meal plan
  Percentage of patients retained in the study

SECONDARY OUTCOMES:
All cause mortality | 6 months follow up period
  Percentage of patients died
Rehospitalization | 6 months follow up period
  Percentage of patients rehospitalized
Emergency room visits | 6 months follow up period
  Percentage of patients visited emergency room
NT-proBNP | 6months follow up period
  Concentration in pg/ml
Kansas City Cardiomyopathy Questionnaire | 6 months follow up period
  The 23-item Kansas City Cardiomyopathy Questionnaire (KCCQ) measures health status in patients with heart failure (HF),
  KCCQ has 6 domains and 2 summary scores:
  Symptom Domain: frequency and burden of symptoms. Physical Function Domain: limitations. Quality of Life (QoL) Domain: reflects QoL Social Limitation Domain: ability to interact in social activities. Self-efficacy Domain: patients' perceptions of how to prevent HF exacerbations. Symptom Stability Domain: recent changes in symptoms. Clinical Summary Score includes total symptom and physical function. Overall Summary Score includes the total symptom, physical function, social limitations and QoL scores.
  The KCCQ is scored by assigning each response an ordinal value, beginning with 1. Scale scores are transformed to a 0 to 100 range by subtracting the lowest possible scale score, dividing by the range of the scale and multiplying by 100. Best is 100.
Food Palatability Questionnaire | 6 months follow up period
  Likert Scales for appearance, taste, and quantity of food (from 1 to 5 - 5 being the most acceptable)

OTHER OUTCOMES:
Systolic Blood Pressure | 6 month follow up
  'mmHg'
Creatinine | 6 month follow up
  'mg/dl'
Blood Urea Nitrogen | 6 month follow up
  'mg/dl'

CONTACTS AND LOCATIONS:
Overall Officials: Javed Butler, MD, MPH, MBA, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalogeropoulos A, Papadimitriou L, Georgiopoulou VV, Dunbar SB, Skopicki H, Butler J. Low- Versus Moderate-Sodium Diet in Patients With Recent Hospitalization for Heart Failure: The PROHIBIT (Prevent Adverse Outcomes in Heart Failure by Limiting Sodium) Pilot Study. Circ Heart Fail. 2020 Jan;13(1):e006389. doi: 10.1161/CIRCHEARTFAILURE.119.006389. Epub 2020 Jan 21. PMID 31959014